CLINICAL TRIAL: NCT00407238
Title: Comparison of Human Corneal Barrier Function With Three Marketed Multi-Purpose Solutions
Brief Title: Corneal Barrier Function With Multi-Purpose Solutions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Collaborators: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 6-08
Record Dates: First submitted 2006-11-17; First posted 2006-12-04 (Estimated); Last update posted 2007-10-23 (Estimated); Status verified 2007-10

CONDITIONS: Contact Lens Care
Keywords: barrier function, multi-purpose solutions, silicone hydrogel contact lenses

INTERVENTIONS:
Device: Multi-purpose solutions (polyquaternium-1 and PHMB)

SUMMARY:
The purpose of this study is to evaluate the effect on epithelial barrier function of three emarketed multi-purpose solution applied to the human eye with hydrogel lenses as during normal regimen use.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect on epithelial barrier function of three emarketed multi-purpose solution applied to the human eye with hydrogel lenses as during normal regimen use.

ELIGIBILITY:
Inclusion Criteria:

* Adapted daily soft contact lens wearers, at least 18 years of age, vision correctable to 20/40

Exclusion Criteria:

* Ocular or systemic allergies, abnormalities of the cornea, active ocular infection, prior keratorefractive surgery, use of ocular medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2006-11; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Ratio of fluorescein dye penetration rate of test eye vs. control

SECONDARY OUTCOMES:
Corneal fluorescein staining

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Paugh, OD, PhD, Principal Investigator — Southern California College of Optometry at Marshall B. Ketchum University
Locations (1):
- Southern California College of Optometry, Fullerton, California, United States